CLINICAL TRIAL: NCT05586776
Title: Decolonization to Reduce After-Surgery Events of Surgical Site Infection
Acronym: DECREASE SSI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Davis (Other); University of California, San Francisco (Other); University of Massachusetts, Amherst (Other); Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Susan Huang, Professor, Division of Infectious Diseases and Medical Director, Epidemiology and Infection Prevention, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1304
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Surgical Site Infection
Keywords: Surgical Site Infection; SSI
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate; Mupirocin; Soaps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Decolonization (Active Comparator): Participants randomized into this arm will perform decolonization using topical antiseptic soap (chlorhexidine body wash) and an antibiotic ointment (nasal mupirocin).
  Interventions: Drug: 4% Chlorhexidine Gluconate; Drug: 2% Mupirocin
- Routine Care (Placebo Comparator): Participants randomized into this arm will perform routine care using soap without antiseptic properties (placebo) and placebo nasal ointment.
  Interventions: Drug: Soap Without Antiseptic Properties (Placebo); Drug: Placebo Nasal Ointment

INTERVENTIONS:
Drug: 4% Chlorhexidine Gluconate — Used for daily showering/bathing for 30 days after hospital discharge.
  Arms: Decolonization
Drug: 2% Mupirocin — Applied to each nostril twice daily for five days for the first two weeks after hospital discharge.
  Arms: Decolonization
Drug: Soap Without Antiseptic Properties (Placebo) — Used for daily showering/bathing for 30 days after hospital discharge.
  Arms: Routine Care
Drug: Placebo Nasal Ointment — Applied to each nostril twice daily for five days for the first two weeks after hospital discharge.
  Arms: Routine Care

SUMMARY:
The DECREASE SSI Trial (Decolonization to Reduce After-Surgery Events of Surgical Site Infection) is a two-arm multi-center individual placebo-controlled randomized (2,700 participants randomized 1:1) clinical trial to reduce post-discharge surgical site infection following open colon or small bowel surgery by comparing chlorhexidine bathing plus nasal mupirocin in the 30 days following discharge to soap without antiseptic properties (placebo) and placebo nasal ointment. This trial seeks to enhance the care of the 675,000 patients annually who undergo colon and small bowel surgery by finding simple and efficacious interventions to reduce SSI.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Recent open (not solely laparoscopic) surgery involving an abdominal incision within the past 14 days. For cesarean section, recruitment restricted to BMI ≥ 40.
* Able to communicate regularly by phone
* Able to bathe, shower or have this task performed by a caregiver

Exclusion Criteria:

* Transfer to an acute care hospital
* Discharged to receive end-of-life hospice measures
* Discharged more than 14 days after surgery
* Allergic to mupirocin and/or chlorhexidine
* Active infection at enrollment*

  *Refers to
  1. Infections requiring systemic antibacterial agents, so viral illness (e.g., COVID, flu) is not an exclusion.
  2. Topical antibacterial agents do not count toward exclusion (e.g., topical products for acne)
  3. Prophylactic antibacterial agents do not count toward exclusion
* Surgical incision not closed at discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to First Post-Discharge Surgical Site Infection | Within 30 Days of Hospital Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Susan Huang, MD, MPH, Principal Investigator — University of California, Irvine; Deborah Yokoe, MD, MPH, Study Director — University of California, San Francisco; Stuart Cohen, MD, Study Director — University of California, Davis
Locations (4):
- United States (4):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California, Irvine Medical Center, Orange, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of California, San Francisco Medical Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
A data request form will be provided to any researcher requesting data from the DECREASE SSI trial This data request form will request the hypothesis/goal of the research, the planned use of the data, and the requested data elements (deidentified only). Any data provided will include the stipulation that use is limited to research purposes only. Requests will not be granted for pursuits directly specified in the grant. If the data request overlaps with additional ongoing post-grant pursuits either by this team or another investigative team that requested the data for a given purpose, a discussion will be pursued toward the potential for joint collaboration.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3 years from publication
Access Criteria: Pending